CLINICAL TRIAL: NCT00000501
Title: Hypertension Prevention Trial (HPT) Feasibility Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 20; R01HL026585-07 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity; Vascular Diseases | interventions — Diet, Sodium-Restricted; Diet, Reducing; Potassium

INTERVENTIONS:
Behavioral: diet, sodium-restricted
Behavioral: diet, reducing
Drug: potassium

SUMMARY:
To test the feasibility and the efficacy of nutritional interventions in the primary prevention of hypertension in individuals predisposed to the development of hypertension; specifically, to test the hypothesis that reduction of weight and/or decreased sodium intake in obese individuals, or decreased sodium intake with or without increased potassium intake (in men and women, regardless of weight) would prevent the elevation of blood pressure and the incidence of hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

The nature of essential hypertension as a mass public health problem throughout the United States, and internationally as well, is recognized generally. Prevalence estimates exceed l5 percent in most adult populations. Further, the results of the Hypertension Detection and Follow-up Program (HDFP) demonstrated the efficacy of antihypertensive therapy even at the 90-l05 mmHg level, which comprises 72 percent of the total hypertensive population. The Joint National Committee on the Detection, Evaluation and Treatment of High Blood Pressure recommended treatment of mild hypertension by pharmacologic or non-pharmacologic therapy to the lowest diastolic pressure consistent with safety and tolerance. The recommendation was consonant with the goal blood pressure guidelines for those with baseline pressures from 90-99 mmHg. Hence, there appeared to be a growing consensus that reduction of blood pressure to levels as low as 80 mmHg might be desirable for optimal cardiovascular health. The Joint National Committee further recommended that, in young patients with uncomplicated mild hypertension, the benefits from pharmacologic therapy must be weighed against the cost, inconvenience, and possible side effects. There was, therefore, a growing concern over the need for pharmacologic management of hypertension and the public health implications of such a course of action. These recommendations toward intervention in mild hypertension set a firm basis for the primary prevention of hypertension.

The association between obesity and elevated blood pressure was widely recognized. Among hypertensive individuals, numerous studies had shown that short term weight reduction by caloric restriction resulted in a reduction of blood pressure. Results of several reports of long-term follow-up of weight reduction efforts indicated that long-term control of weight at levels compatible with the objectives of the HPT was feasible. A number of investigators had achieved these levels one or more years after treatment despite minimal intervention efforts during the follow-up period.

There was strong circumstantial evidence relating sodium intake to hypertension. Most impressive evidence came from the study of the 'low-salt tribes', subsisting on a very low sodium intake. They failed to develop hypertension, or even gradual rise of blood pressure with age. Many studies published on the effect of lowering sodium intake on blood pressure of hypertensive patients had been positive. In one investigation, blood pressure fell approximately 9 (systolic)/6 (diastolic) mmHg when sodium intake was reduced from approximately l80 to l00 mEq/day. Reduction of sodium intake to a level of 70-l00 mEq/day appeared within the capability of most people and maintenance up to a period of two years had been indicated with minimal follow-up procedures.

The role of potassium intake in the development and treatment of hypertension was less clear. As noted above, primitive cultures studied epidemiologically had low sodium intakes associated with low prevalence and incidence of hypertension but these cultures also consumed higher levels of potassium. It has been suggested that the ratio of sodium to potassium may be the most important determinant of blood pressure. Hygienic intervention to increase potassium intake in free-living populations was the least studied of the procedures used in the HPT. Potassium intakes > l00 mEq could be achieved without the use of dietary supplements if individuals consumed large quantities of fruits and vegetables. This natural intake could also be increased by use of potassium-based baking powder and seasonings.

The study was carried out by four clinical and two resource centers (a Coordinating Center and a Nutrition and Educational Resource Center). It was to be Phase l of a long-term intervention trial to determine whether development of hypertension could be prevented in a population at special risk. The initial phase of the study was directed towards testing the feasibility of the intervention, alternative modes of recruitment, quantification of sodium and potassium intake, trends in blood pressure, and the pre-testing of various study procedures.

Each of the four clinical centers recruited 200 or more eligible 25 to 49 year old individuals (total 841), either identified through any of a number of multiple community sources, or through an index of hypertensive cases. The clinical investigators aided by statistical and data processing support from the Data Coordinating Center and intervention support through a special Nutrition and Education Resources Center, formed the collaborative group to test the working hypothesis. The study protocol was completed in the fall of 1982. Recruitment ended September 30, 1983. The three-year follow-up period ended August 1986. Analysis of the data ended in December 1988.

DESIGN NARRATIVE:

A randomized, non-blind design with three treatment groups (non-obese) or five groups (obese), including a no-treatment group in each weight stratum. Intervention methods were dietary only, and included sodium restriction, sodium restriction plus potassium supplementation (obese and non-obese), weight reduction, and weight reduction plus sodium restriction (obese only). This was a pilot study with measures of feasibility including recruitment success, dietary adherence, and blood pressure differences among the treatment groups.

ELIGIBILITY:
Men and women, ages 25 to 49. Diastolic blood pressure between 78 and 89 mm Hg. Free of major disease. Not on a special diet or antihypertensive medication at entry. Some mild to moderately obese subjects.

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1981-09; Study Completion 1986-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nemat Borhani — University of California, Davis; Robert Jeffery — University of Minnesota; Herbert Langford — University of Mississippi Medical Center; Albert Oberman — University of Alabama at Birmingham; Ronald Prineas — University of Minnesota

REFERENCES:
- [Background] Hypertension Prevention Trial Research Group: Hypertension Prevention Trial--First Year Dietary Changes. In Strasser T, Ganten D, (Eds.). Mild Hypertension: From Drug Trials to Practice, New York, Raven Press, 1987.
- [Background] Meinert CL, Borhani NO, Langford HG. Design, methods, and rationale in the Hypertension Prevention Trial. Hypertension Prevention Trial Research Group. Control Clin Trials. 1989 Sep;10(3 Suppl):1S-29S. doi: 10.1016/0197-2456(89)90040-8. PMID 2680271
- [Background] Borhani NO, Tonascia J, Schlundt DG, Prineas RJ, Jefferys JL. Recruitment in the Hypertension Prevention trial. Hypertension Prevention Trial Research Group. Control Clin Trials. 1989 Sep;10(3 Suppl):30S-39S. doi: 10.1016/0197-2456(89)90041-x. PMID 2680272
- [Background] Brown KM, Oberman A, Van Natta ML, Forster JL. Baseline characteristics in the Hypertension Prevention Trial. Hypertension Prevention Trial Research Group. Control Clin Trials. 1989 Sep;10(3 Suppl):40S-64S. doi: 10.1016/0197-2456(89)90042-1. PMID 2680273
- [Background] Jeffery RW, Tonascia S, Bjornson-Benson W, Schlundt DG, Sugars C. Treatment in the Hypertension Prevention Trial. Hypertension Prevention Trial Research Group. Control Clin Trials. 1989 Sep;10(3 Suppl):65S-83S. doi: 10.1016/0197-2456(89)90043-3. PMID 2680274
- [Background] Prud'homme GJ, Canner PL, Cutler JA. Quality assurance and monitoring in the Hypertension Prevention Trial. Hypertension Prevention Trial Research Group. Control Clin Trials. 1989 Sep;10(3 Suppl):84S-94S. doi: 10.1016/0197-2456(89)90044-5. PMID 2680275
- [Background] Tonascia J, Donithan M, Tonascia S, et al for the Hypertension Prevention Trial Research Group: Hypertension Prevention Trial: Estimation of 24-hour Sodium and Potassium Excretion from Overnight Urine Collections. Baltimore, Maryland, Department of Biostatistics, Johns Hopkins University, Technical Report 703, 1989.
- [Background] Shah M, Jeffery RW, Hannan PJ, Onstad L. Relationship between socio-demographic and behaviour variables, and body mass index in a population with high-normal blood pressure: Hypertension Prevention Trial. Eur J Clin Nutr. 1989 Sep;43(9):583-96. PMID 2606089
- [Background] The Hypertension Prevention Trial: three-year effects of dietary changes on blood pressure. Hypertension Prevention Trial Research Group. Arch Intern Med. 1990 Jan;150(1):153-62. PMID 2404477
- [Background] Jeffery RW, French SA, Schmid TL. Attributions for dietary failures: problems reported by participants in the Hypertension Prevention Trial. Health Psychol. 1990;9(3):315-29. doi: 10.1037//0278-6133.9.3.315. PMID 2187695
- [Background] Forster JL, Jeffery RW, VanNatta M, Pirie P. Hypertension prevention trial: do 24-h food records capture usual eating behavior in a dietary change study? Am J Clin Nutr. 1990 Feb;51(2):253-7. doi: 10.1093/ajcn/51.2.253. PMID 2407098
- [Background] Shah M, Jeffery RW, Laing B, Savre SG, Van Natta M, Strickland D. Hypertension Prevention Trial (HPT): food pattern changes resulting from intervention on sodium, potassium, and energy intake. Hypertension Prevention Trial Research Group. J Am Diet Assoc. 1990 Jan;90(1):69-76. PMID 2404050
- [Background] Schmid TL, Jeffery RW, Onstad L, Corrigan SA. Demographic, knowledge, physiological, and behavioral variables as predictors of compliance with dietary treatment goals in hypertension. Addict Behav. 1991;16(3-4):151-60. doi: 10.1016/0306-4603(91)90007-5. PMID 2063702
- [Background] Canner PL, Borhani NO, Oberman A, Cutler J, Prineas RJ, Langford H, Hooper FJ. The Hypertension Prevention Trial: assessment of the quality of blood pressure measurements. Am J Epidemiol. 1991 Aug 15;134(4):379-92. doi: 10.1093/oxfordjournals.aje.a116100. PMID 1877599